CLINICAL TRIAL: NCT03284463
Title: Safety and Efficacy of Glibenclamide Combined With Rt-PA in Treating Acute Ischemic Stroke: a Prospective, Randomized, Double-blind, Placebo-control, Multi-center Study
Brief Title: Safety and Efficacy of Glibenclamide Combined With Rt-PA in Acute Cerebral Embolism
Acronym: SE-GRACE
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NFEC-2017-130
Record Dates: First submitted 2017-09-14; First posted 2017-09-15 (Actual); Last update posted 2023-06-12 (Actual); Status verified 2023-06

CONDITIONS: Acute Stroke
Keywords: acute ischemic stroke; glibenclamide; rt-PA; blood-brain barrier; brain edema
MeSH Terms: conditions — Stroke; Ischemic Stroke; Brain Edema | interventions — Glyburide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Glibenclamide (Active Comparator): Glibenclamide Tablets
  Interventions: Drug: Glibenclamide
- Placebo (Placebo Comparator): Placebo for Glibenclamide
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Glibenclamide — Glibenclamide is administered with a loading dose of 1.25 mg within 10 hours of stroke onset, orally or through gastric tube, followed by 0.625 mg every 8 hour for 5 days.
  Arms: Glibenclamide
Drug: Placebo — Placebo is administered with a loading dose of 1.25 mg within 10 hours of stroke onset, orally or through gastric tube, followed by 0.625 mg every 8 hour for 5 days.
  Arms: Placebo

SUMMARY:
This study is designed to evaluate the safety and efficacy of oral glibenclamide in acute ischemic stroke patients who under intravenous rt-PA thrombolysis.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of acute ischemic stroke in the MCA territory (PCA and/or ACA territory involvement in addition to primary MCA territory stroke is acceptable)
* Aged ≥18 and ≤74 years
* A baseline NIHSS score between 4 to 25
* Intravenous rt-PA thrombolysis conducted within 4.5 hours after stroke onset, if known, or the time last seen well [termed "time last known at neurologic baseline" (TLK@B)]
* The time to the start of administration of Study Drug must be ≤10 h after time of symptom onset or TLK@B
* Informed consent was signed by the subject or the legal representative

Exclusion Criteria:

* Prior to stroke, significant disability exists, with modified Rankin Scale >1 point
* With medical history or evidence of cerebral hemorrhage, subarachnoid hemorrhage, arteriovenous malformation, cerebral aneurysm or brain tumor
* With clinical or imaging evidence of contralateral cerebral infarction which is believed to have influence on the patient outcome by the investigators
* With clinical or imaging evidence of occlusion in vertebral or basilar artery
* With clinical evidence of brain herniation, e.g., one or two dilated, fixed pupils; unconsciousness (i.e., C2 on item 1a on the NIHSS); and/or loss of other brainstem reflexes, attributable to edema or herniation according to the investigator's judgment
* With gastrointestinal bleeding and instable hemodynamics or other causes that force the patient to stop nutritional support
* Renal disorder from the patient's history (e.g., dialysis) or eGFR of <60 mL/min/1.73 m2
* Severe liver disease, or ALT >3 times upper limit of normal or bilirubin >2 times normal (subjects may be randomized if liver function tests have been drawn but are not yet available and the subject has no known history of liver disease; however treatment with Study Drug cannot commence until liver function tests are available and indicate ALT >3 times upper limit of normal and bilirubin >2 times upper limit of normal)
* Blood glucose <3.0 mmol/L at enrollment or immediately prior to administration of Study Drug, or a clinically significant history of hypoglycemia
* Acute ST elevation myocardial infarction, and/or acute decompensated heart failure, and/or Tc > 520 ms, and/or known history of cardiac arrest (PEA, VT, VF, asystole), and/or admission for an acute coronary syndrome, myocardial infarction, or coronary intervention within the past 3 months
* Known sulfonylurea treatment within 7 days. Sulfonylureas include glyburide/glibenclamide; glibenclamide plus metformin; Xiaoke Pill (a Chinese patent medicine with main effective constituent of glibenclamide); glimepiride; repaglinide; nateglinide; glipizide; gliclazide; tolbutamide; glibornuride
* Known treatment with bosentan within 7 days
* Known allergy to sulfa or specific allergy to sulfonylurea drugs
* Known G6PD enzyme deficiency
* Pregnant women. Women must be either postmenopausal (as confirmed by the LAR), permanently sterilized or, if ≤50 years old must have a negative test for pregnancy obtained before enrollment
* Breast-feeding women who do not agree (or their LAR does not agree) to stop breastfeeding during Study Drug infusion and for 7 days following the end of Study Drug infusion
* Patients already enrolled in a non-observation-only stroke study, or with life-expectancy <6 months not related to current stroke, or those unlikely to be compliant with follow up
* Patients currently receiving an investigational drug
* Mentally incompetent (prior to qualifying stroke) patients and wards of the state
* Patients who, in the opinion of the investigator, are not suitable for the study (reason to be documented)

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 306 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2022-08-28 (Actual); Study Completion 2023-05-28 (Actual)

PRIMARY OUTCOMES:
Functional outcome: The proportion of mordified Rankin Scale of 0 to 2 points | 90 days after the stroke onset
  The proportion of mordified Rankin Scale of 0 to 2 points at 90 days

SECONDARY OUTCOMES:
Early improvement: The proportion of NIHSS decreased ≥ 4 points | 7 days after the stroke onset
  The proportion of NIHSS decreased ≥ 4 points at 7 days
Hemorrhagic transformation: The proportion of parenchymal hemorrhagic transformation in cranial CT | 96 hours after the stroke onset
  The proportion of parenchymal hemorrhagic transformation in cranial CT within 96 hours
Midline shift: The proportion of midline shift ≥ 6 mm in cranial CT | 96 hours after the stroke onset
  The proportion of midline shift ≥ 6 mm in cranial CT within 96 hours
Functional outcome 2: The modified Rankin Scale distribution | 90 days after the stroke onset
  The modified Rankin Scale distribution at 90 days
Functional outcome 3: The proportion of Barthel Index of 60-100 points | 90 days after the stroke onset
  The proportion of Barthel Index of 60-100 points
Functional outcome 4: The proportion of IQCODE of ≤ 3.40 | 6 months and 1 year after the stroke onset
  The proportion of Informant Questionnaire on Cognitive Decline in the Elderly (IQCODE) of ≤ 3.40 at 6 months and 1 year after the stroke onset
Blood-brain barrier: The serum concentration of MMP-9 | Baseline, 24, 48, and 72 hours after the stroke onset
  The serum concentration of MMP-9 at baseline, and at 24, 48, and 72 h

OTHER OUTCOMES:
Mortality | 90 days after the stroke onset
  The mortality at 90 days
Early neurological deterioration | 24 hours after the stroke onset
  The ratio of neurological deterioration (NIHSS increased ≥ 4 points) within 24 hours after the onset
Hypoglycemia | 5 days after the stroke onset
  The incidence of hypoglycemia (random blood glucose < 3.9 mmol/L)
Cardiac events | 30 days after the stroke onset
  The incidence of cardiac events in cardiac examination (ECG, echocardiography)
Pulmonary infection | 7 days within the stroke onset
  The incidence of pulmonary infection
AEs and SAEs | 30 days after the stroke onset
  The incidence of adverse event and serious adverse event

CONTACTS AND LOCATIONS:
Overall Officials: Suyue Pan, M.D., Ph.D., Principal Investigator — Department of Neurology, Nanfang Hospital, Southern Medical University
Locations (8):
- China (8):
  - Huadu District People's Hospital of Guangzhou, Guangzhou, Guangdong
  - Nanfang Hospital of Southern Medical University, Guangzhou, Guangdong
  - Heyuan People's Hospital, Heyuan, Guangdong
  - Maoming People's Hospital, Maoming, Guangdong
  - Maoming Traditional Chinese Medical Hospital, Maoming, Guangdong
  - Hainan Provincial Hospital of Traditional Chinese Medicine, Haikou, Hainan
  - Haikou People's Hospital, Haikou, Hainan
  - The First Affiliated Hospital of Wenzhou Medical University, Wenzhou, Jiangsu

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Huang K, Zhao X, Zhao Y, Yang G, Zhou S, Yang Z, Huang W, Weng G, Chen P, Duan C, Lin Z, Wang S, Liu X, Huang Y, Zhang J, Zhang X, Li H, Ye S, Gu Y, Zhu M, Chen W, Quan W, Liu N, Chen Q, Chang Y, He J, Ji Z, Wu Y, Pan S; SE-GRACE Collaborators. Safety and efficacy of glibenclamide combined with rtPA in acute cerebral ischemia with occlusion/stenosis of anterior circulation (SE-GRACE): a randomized, double-blind, placebo-controlled trial. EClinicalMedicine. 2023 Nov 1;65:102305. doi: 10.1016/j.eclinm.2023.102305. eCollection 2023 Nov. PMID 37965431
- [Derived] Huang K, Ji Z, Wu Y, Huang Y, Li G, Zhou S, Yang Z, Huang W, Yang G, Weng G, Chen P, Pan S. Safety and efficacy of glibenclamide combined with rtPA in acute cerebral ischemia with occlusion/stenosis of anterior circulation (SE-GRACE): study protocol for a randomized controlled trial. BMC Neurol. 2020 Jun 11;20(1):239. doi: 10.1186/s12883-020-01823-z. PMID 32527232